CLINICAL TRIAL: NCT01309581
Title: Ketamine Anesthesia to Enhance Efficacy and Tolerability of Electroconvulsive Therapy in Patients With Unipolar or Bipolar Depression
Brief Title: Use of Ketamine to Enhance Electroconvulsive Therapy (ECT) in Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: limited enrollment
Sponsor: James Murrough (Other)
Responsible Party: Sponsor-Investigator, James Murrough, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 09-2251; KETECT-MSSM-01
Record Dates: First submitted 2011-03-02; First posted 2011-03-07 (Estimated); Results first posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-07

CONDITIONS: Major Depression; Bipolar Depression
Keywords: depression; electroconvulsive therapy; ketamine; antidepressant
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Depression | interventions — Ketamine; Methohexital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): Participants receiving ECT for depression will be randomized 1:1 to either ketamine (experimental condition) or methohexital (standard anesthetic).
  Interventions: Drug: Ketamine
- Methohexital (Active Comparator): Participants receiving ECT for depression will be randomized 1:1 to either ketamine (experimental condition) or methohexital (standard anesthetic).
  Interventions: Drug: Methohexital

INTERVENTIONS:
Drug: Ketamine — Ketamine 1-2 mg/kg IV as indicated for ECT
  Arms: Ketamine
Drug: Methohexital — Methohexital 1 mg/kg IV as indicated for ECT
  Arms: Methohexital

SUMMARY:
The primary objectives of this study are to investigate the potential for ketamine anesthesia to increase the antidepressant efficacy of Electroconvulsive therapy (ECT) and to decrease acute ECT-induced adverse cognitive effects.

DETAILED DESCRIPTION:
Electroconvulsive therapy (ECT) is one of the most robust antidepressant treatments available. However, there is the potential for significant acute and longer term adverse cognitive effects with ECT and the antidepressant response requires multiple treatment sessions, increasing risk of adverse effects. Further, antidepressant response to ECT is often less than maximal and relapse is common. Growing preclinical and clinical evidence of the rapid-acting antidepressant properties of the anesthetic agent ketamine suggests the use of ketamine anesthesia as a strategy to increase rate of response and shorten treatment course in the administration of ECT. In addition, preclinical and clinical evidence suggests the potential of ketamine to decrease the adverse cognitive effects associated with ECT.

The investigators propose a pilot study to measure both acute therapeutic efficacy and cognitive side effects of ECT using ketamine compared to methohexital in depressed patients. The investigators will also explore other parameters of ECT such as seizure duration and morphology, as well as hemodynamic and behavioral changes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients: 18 to 59 years
2. Women of childbearing potential must agree to use a medically accepted means of contraception for the duration of the study
3. DSM IV MINI diagnosis of major depressive episode (MDD), unipolar or bipolar
4. Pretreatment 24-item Hamilton Rating Scale for Depression score > 21
5. ECT is clinically indicated
6. Patient has the capacity to provide informed consent.

Exclusion Criteria:

1. DSM-IV diagnosis of schizophrenia, schizoaffective disorder, or mental retardation
2. Current primary diagnosis of anxiety disorder, obsessive- compulsive disorder, or eating disorder that precedes the onset of the current episode of depression
3. Current diagnosis of delirium, dementia, or amnestic disorder
4. Baseline Mini Mental State Exam (MMSE) score < 24 and a total score falling two standard deviations below the age- and education-adjusted mean
5. Any active general medical condition or CNS disease which can affect cognition or response to treatment
6. Current (within the past three months) diagnosis of active substance dependence, or active substance abuse within the past week
7. Lifetime history of ketamine or PCP abuse or dependence
8. ECT within three months
9. The presence of any known or suspected contraindication to methohexital or ketamine including but not limited to known allergic reactions to these agents, uncontrolled hypertension arrhythmia severe coronary artery disease and porphyria
10. Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James W Murrough, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine | Methohexital
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Methohexital | Total
Number analyzed (Participants) | 2 | 1 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 53 (5.6) | 50 (0) | 50 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression-24 (HRSD24)
Description: The HDRS-24 is used to rate depressive symptoms. This instrument is considered one of the "gold standard" clinician-rated instruments for depressive symptoms. We have established procedures for the maintenance of inter-rater reliability.
Time Frame: Change from beginning of ECT treatment to end; on average 3 weeks
Arm/Group | Ketamine | Methohexital
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Quick Inventory of Depressive Symptomatology, Self Report (QIDS-SR)
Description: The QIDS-SR is a 16-item self-rated instrument designed to assess the severity of depressive symptoms present in the past seven days (Rush et al 2003). The 16 items cover the nine symptom domains of major depression, and are rated on a scale of 0-3. Total score ranges from 0 to 27, with ranges of 0-5 (normal), 6-10 (mild), 11-15 (moderate), 16-20 (moderate to severe), and 21+ (severe).
Time Frame: Change from beginning of ECT treatment to end; on average 3 weeks
Arm/Group | Ketamine | Methohexital
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ketamine | Methohexitol
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=2) | Methohexitol (N=1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Frequent Urination (Renal and urinary disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness on standing (Cardiac disorders) | 1 (1) | 0 (0)
Sleep disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Restlessness (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination, limited enrollment, data analysis not done due to technical problems with measurement leading to unreliable and uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No